CLINICAL TRIAL: NCT05850871
Title: Evaluation of Ceftazidime-avibactam Plus Aztreonam in Patients Infected by MBL-producing Enterobacterales and CRISPR/Cas9-based Strategy for Curing Drug-resistant Genes
Brief Title: Drug Resistance Mechanism of Enterobacteriaceae and Its Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Mingju Hao, Clinical Professor, Qianfoshan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: JNQH-CT-231001
Record Dates: First submitted 2023-04-06; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection
Keywords: carbapenem resistance; Enterobacteriaceae; CRISPR/Cas9
MeSH Terms: interventions — Aztreonam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAZ/AVI plus Aztreonam (Experimental): CAZ-AVI was administered at the dose of 2.5 g every 8 hours and ATM at the dose of 2 g every 8 hours
  Interventions: Drug: CAZ/AVI plus Aztreonam
- Conventional treatment (Active Comparator): Other active antibiotics were administered, including colistin, tigecycline, fosfomycin, meropenem.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Drug: CAZ/AVI plus Aztreonam — Samples of the patients will be examined such as the routine blood test, blood culture et al.
  Other Names: ceftzadime avibactam, aztreonam
  Arms: CAZ/AVI plus Aztreonam
Other: Conventional treatment — Conventional treatment
  Arms: Conventional treatment

SUMMARY:
The first aim of this study is to explore the drug resistance mechanism of Enterobacteriaceae bacteria and to evaluate the treatment effect of ceftazidime-avibactam (CAZ-AVI) in combination with aztreonam (ATM) against Metallo-β-lactamases (MBL) producing Enterobacterales in vivo. The investigators then use CRISPR/Cas9 technology to remove Enterobacteriaceae bacteria resistance and virulence genes

DETAILED DESCRIPTION:
Clinical information of subjects, including diseases, departments, medication history, days of hospitalization, and treatment outcomes will be collected; Bacterial species names will be identified and drugs sensitivity will be detected; For patients with bloodstream infection of MBL-producing Enterobacterales, ceftazidime-avibactam (CAZ-AVI) was administered at the dose of 2.5 g every 8 hours and aztreonam (ATM) at the dose of 2 g every 8 hours.

The primary outcome measure was 30-day all-cause mortality, while secondary outcomes were clinical failure at day 14 and length of stay (LOS) after bloodstream infection diagnosis. Cox regression analysis, including a propensity score (PS) for receiving CAZ-AVI plus ATM, was conducted to assess the primary and secondary outcomes. The CRISPR/Cas9 gene curation technology was used to eliminate the drug resistance and virulence factors of Enterobacteriaceae in the mouse intestinal colonization model.

ELIGIBILITY:
Inclusion Criteria:

* Subjects clinically suspected of infection caused by Enterobacterales
* Subjects with bloodstream infection by MBL-producing Enterobacterales

Exclusion Criteria:

* Infections caused by viruses, fungi, atypical pathogens, and other non-Enterobacteriaceae bacteria
* subjects who are unwilling to enter the research group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | two years
  The primary outcome measure was 30-day all-cause mortality
clinical failure at day 14 | two years
  severe comorbidities, mechanical ventilation or septic shock at day 14
length of stay after diagnosis | two years
  length of stay (LOS) after blood stream infection diagnosis

SECONDARY OUTCOMES:
Positive rate of Metallo-β-lactamases (MBL) producing Enterobacterales | two years
  Positive rate and subtype distribution of Metallo-β-lactamases (MBL) producing Enterobacterales

OTHER OUTCOMES:
Curation index as assessed by MBL producing Enterobacterales compared with MBL negative Enterobacterales. | two years
  Evaluation of the efficienty of CRISPR/Cas9 technique to cure resistance genes in a mouse model colonized by multidrug resistant enterobacteriaceae. Curation index as assessed by MBL producing Enterobacterales compared with MBL negative Enterobacterales isolated from the feces sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jiasheng Zhang, Doctor, Study Director — Shandong First Medical University
Locations (1):
- Mingju Hao, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No